CLINICAL TRIAL: NCT06773286
Title: Establishing the Feasibility, Safety, and Efficacy of Spinal Cord Transcutaneous Stimulation with Activity-based Training for Upper Extremity Function Recovery in Individuals with Acute to Subacute Tetraplegia
Brief Title: Combining Spinal Cord Transcutaneous Stimulation and Activity-based Training in Inpatient Rehabilitation to Facilitate Upper Limb Function of Individuals with Acute to Subacute Cervical Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Fan Zhang, Principal Investigator, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 40652; CSCR23ERG001 (Other Grant/Funding Number: NEW JERSEY COMMISSION ON SPINAL CORD RESEARCH)
Record Dates: First submitted 2025-01-02; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Spinal Cord Injury Cervical
Keywords: Spinal Cord Injury; Inpatient Rehabilitation; Upper Extremity; Spinal Cord Transcutaneous Stimulation; Activity-based Training
MeSH Terms: conditions — Spinal Cord Injuries | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active Spinal Cord Transcutaneous Stimulation Combined with Activity-based Training (Active Comparator): Participants will receive activity-based training (ABT) while receiving concomitant, active spinal stimulation (scTS) applied at the cervical and thoracic spinal segments over the dorsal skin with optimized and customized stimulation parameters. Round self-adhesive electrodes will be placed over the skin at the midline of spinous processes as cathodes and a pair of rectangular anodes electrodes will be placed over the anterior iliac crests of the pelvis. The stimulation waveform is rectangular pulse with 1-ms duration filled with a carrier frequency of 5kHz. Target simulation will be sub-threshold for UE muscle activation and verified by the absence of visible muscle contraction. The stimulation parameters will be adjusted as needed throughout the intervention course based on the participant's performance and comfort level. The intervention will be administered over 2 consecutive weeks, for 30mins/session and 5 sessions/week, as a part of their daily 3-hour therapy.
  Interventions: Other: Active Stimulation
- Sham Spinal Cord Transcutaneous Stimulation Combined with Activity-based Training (Sham Comparator): The sham-control group will go through ABT paired with sham stimulation to control for placebo effects associated with the perception of scTS. Stimulation will be delivered at one cervical location. No stimulation mapping procedure will be performed. During the training session, the stimulation intensity will be briefly ramped up to a level at which the participants report perceiving the stimulation, and then ramped down to 0mA at both the start and the end of session. The stimulator and electrodes will remain attached to the participant while receiving ABT training. The intervention will be administered over 2 consecutive weeks, for 30mins/session and 5 sessions/week, as a part of their daily 3-hour therapy.
  Interventions: Other: Sham
- Activity-based Training Only (Other): Participants in ABT group will receive ABT only. ABT will concentrate on activities of gross UE movement, grasping, pinching, gross and fine motor skill. The hand grasp task will focus on grasping objects with different shapes and weights (i.e. weighted container and tennis ball) and placing/removing them from small storage container; the pinch task involves picking up, translating, and releasing small objects with varied sizes (i.e. blocks, dices, marble balls, nuts, etc.). The training therapist selects tasks based on participant's level of impairment and individual goals. The dosage of ABT will be 30 minutes/session, with approximately 15 minutes allocated on each side.
  Interventions: Other: Training only

INTERVENTIONS:
Other: Active Stimulation — Participants will receive activity-based training (ABT) while receiving concomitant, active spinal stimulation (scTS) applied at the cervical and thoracic spinal segments over the dorsal skin with optimized and customized stimulation parameters. Round self-adhesive electrodes will be placed over the skin at the midline of spinous processes as cathodes and a pair of rectangular anodes electrodes will be placed over the anterior iliac crests of the pelvis. The stimulation waveform is rectangular pulse with 1-ms duration filled with a carrier frequency of 5kHz. Target simulation will be sub-threshold for UE muscle activation and verified by the absence of visible muscle contraction. The stimulation parameters will be adjusted as needed throughout the intervention course based on the participant's performance and comfort level. The intervention will be administered over 2 consecutive weeks, for 30mins/session and 5 sessions/week, as a part of their daily 3-hour therapy.
  Arms: Active Spinal Cord Transcutaneous Stimulation Combined with Activity-based Training
Other: Sham — The sham-control group will go through ABT paired with sham stimulation to control for placebo effects associated with the perception of scTS. Stimulation will be delivered at one cervical location. No stimulation mapping procedure will be performed. During the training session, the stimulation intensity will be briefly ramped up to a level at which the participants report perceiving the stimulation, and then ramped down to 0mA at both the start and the end of session. The stimulator and electrodes will remain attached to the participant while receiving ABT training. The intervention will be administered over 2 consecutive weeks, for 30mins/session and 5 sessions/week, as a part of their daily 3-hour therapy.
  Arms: Sham Spinal Cord Transcutaneous Stimulation Combined with Activity-based Training
Other: Training only — articipants in ABT group will receive ABT only. ABT will concentrate on activities of gross UE movement, grasping, pinching, gross and fine motor skill. The hand grasp task will focus on grasping objects with different shapes and weights (i.e. weighted container and tennis ball) and placing/removing them from small storage container; the pinch task involves picking up, translating, and releasing small objects with varied sizes (i.e. blocks, dices, marble balls, nuts, etc.). The training therapist selects tasks based on participant's level of impairment and individual goals. The dosage of ABT will be 30 minutes/session, with approximately 15 minutes allocated on each side.
  Arms: Activity-based Training Only

SUMMARY:
The purpose of this clinical trial is to understand the safety and practicality of using spinal cord transcutaneous (through the skin) stimulation in an inpatient setting as well as how the combination of activity-based training (ABT) and spinal cord transcutaneous stimulation (scTS) can improve participants' ability to use their hands, arms, and trunk in an inpatient rehabilitation program. The main questions it aims to answer are:

* Is the combination of spinal cord transcutaneous stimulation and ABT is safe and practical when applied to individuals with acute to subacute cervical SCI during inpatient rehabilitation?
* How the combined intervention can improve hand and arm function when applied to those individuals? The investigators will assess the safety, feasibility, and preliminary efficacy of the combined intervention and compare to a sham control (sham stimulation combined with ABT) and a ABT only group to see if the combined intervention can lead to greater function recovery.

Participants will:

* Receive one type of the three intervention (scTS+ABT, sham scTS+ABT, or ABT only) for 10 sessions with 30 mins/session over 2 weeks.
* Receive assessment before, during, and immediately after the intervention, and at 1-month, 2-month, and 3-month follow-up visits.

DETAILED DESCRIPTION:
The objective of this study is to investigate the use of scTS combined with ABT in inpatient rehabilitation, to facilitate UE functional recovery for individuals with acute to subacute cervical SCI. The investigators will assess the safety, feasibility, and preliminary efficacy of the combined intervention with a 10-day regimen in a randomized, sham-controlled clinical trial. The investigators hypothesize that the combination of scTS+ABT applied in individuals with acute to subacute cervical SCI will 1) be both safe and feasible when implemented as a part of the medical care in an inpatient SCI rehabilitation program, and 2) promote greater improvements in UE function compared to sham control and ABT alone. In addition, the investigators will explore the potential neurophysiological mechanism underlying the combined intervention by evaluating the pre-post changes of cortical and spinal excitability. The investigators anticipate that the functional outcome improvements will be associated with the gains of cortical and spinal excitability.

(Aim 1) To determine whether scTS+ABT intervention is safe when applied to persons with acute to subacute cervical SCI during inpatient rehabilitation. The investigators will evaluate the intervention safety based on the adverse event reports focusing three categories: (1) scTS-related (pain/discomfort and skin integrity), (2) ABT-related (musculoskeletal injuries, heart rate, and oxygen saturation levels), and (3) SCI-related (spasticity and autonomic dysreflexia). The type, frequency, and severity of adverse events reported in scTS+ABT group will be compared to those from ABT alone group. (Aim 2) To examine whether a 10-day regimen of scTS+ABT is feasible to apply to individuals with acute to subacute SCI during an inpatient rehabilitation program. The interest and willingness of participants to enroll and complete this study will provide insight into the feasibility of scTS+ABT intervention. The investigators will assess the feasibility based on quantitative data including ease of recruitment (accrual rate) and study completion rate and compare the study completion rate in scTS+ABT and ABT alone group. (Aim 3) To evaluate the efficacy of scTS+ABT intervention in promoting UE functional recovery in acute to subacute SCI, as compared to the sham control and ABT only. Given the greatest opportunity for recovery and neuroplasticity in acute-subacute SCI stage and the promising results demonstrated in the previous chronic SCI studies, the investigators expect that applying scTS+ABT at early stages would lead to greater UE function improvements compared to scTSsham+ABT and ABT only. UE motor impairment, voluntary handgrip strength, and UE functional ability will be quantitatively assessed three time at baseline, once at the end of intervention, and once at 1-, 2-, 3-month follow up. Within-group and between-group comparison will be made to evaluate the efficacy of different interventions. (Aim 4, Exploratory) To quantify and characterize the neurophysiological changes after scTS+ABT, as compared to the sham control or ABT alone. Previous chronic studies have suggested that scTS can increase the excitability of spinal network and activate the motor neurons within spinal cord distal to the lesion, leading to restoration of voluntary motor control. Here, the investigators will examine whether a 10-day regimen of scTS+ABT applied in the acute to subacute stage can also lead to neurophysiological gains. Pre-post changes in the cortical and spinal excitability will be measured and compared to the sham control and ABT only group. As an exploratory aim, the investigators will evaluated on a subset sample of each group (n=4).

ELIGIBILITY:
Inclusion Criteria:

* must be at least 18 years of age.
* must have had a spinal cord injury for less than or equal to 8 weeks.
* must have a traumatic cervical SCI with lesions (AIS A or B, C5-C7).
* must have some degree of motor dysfunction in the hand (bilateral UE motor score <25).
* must be medically stable enough to participate in activity-based recovery training.
* must be able to tolerate spinal cord transcutaneous stimulation, as determined by study staff.
* must have ability to understand and the willingness to sign an informed consent.

Exclusion Criteria:

* have a history of seizures, head trauma and/or cognitive deficit
* have surgically implanted foreign bodies such as a pacemaker, metal plate in the skull, and metal inside the skull
* have a pressure sore or skin issues.
* have severe spasticity.
* in medically unstable condition.
* have a history of illicit drug abuse.
* have a history of medical disorders of my heart, lungs, bladder, kidneys or other parts of my body that are unrelated to my spinal cord injury.
* unable or unwilling to wean from anti-spasticity medication (for an example: baclofen, Xeomin, and Lioresal).
* unable to meet the attendance requirements.
* currently enrolled in another interventional research study.
* unable to follow instructions and maintain alertness during assessments and training.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change of pain before and after daily intervention | From the beginning to the end of each intervention session at 30 minutes
  Subjects will be asked to rate their pain intensity using an 11-point Numerical Rating Scale (i.e. 0-10), before and after each intervention session. The change in pain will be documented.
Change of skin integrity before and after daily intervention session | From the beginning to the end of each intervention session at 30 minutes
  Skin integrity under electrode placement site will be assessed by a clinician before and after each session, any change i.e., redness, swelling, breakdown, will be recorded.
Study completion rate | From enrollment to the post-intervention assessment at 3 weeks
  Study completion rate will be calculated at post-intervention by dividing the number of participants who will be present at these time points by the number of individuals who are enrolled and begin the intervention.

SECONDARY OUTCOMES:
Adverse event after daily intervention session | At the end of each intervention session at 30 minutes
  An adverse events survey will be completed on a daily basis to evaluate adverse effects potentially related to spinal stimulation, activity-based training, and SCI.
Change of Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) Scores | From baseline to the end of intervention at 2 weeks, post-intervention at 1 month, 2 months, and 3 months
  GRASSP is a standard clinical outcome measure used to evaluate the hand and UE function in people with cervical SCI. Specifically, this outcome measure evaluates UE strength, sensation, the ability to complete different grasp patterns, and the ability to utilize those grasp patterns to successfully complete functional activities. It consists of four subtests for each upper limb: dorsal and palmar sensation, strength (tested with motor grading of 10 muscles), and prehension (distinguishes scores for qualitative and quantitative grasping). The numerical scores in each subtest provide a comprehensive assessment of UE function.
Change of voluntary handgrip forces | From baseline to the end of intervention at 2 weeks, post-intervention at 1 month, 2 months, and 3 months
  Maximum voluntary handgrip forces will be measured from both hands by using a hand-held dynamometer (Echo, JTECH Medical, Midvale, Utah) with stimulation turned off. To avoid compensation movement (tenodesis), testing will be performed in a standardized way with participants seated upright, shoulder adducted and neutrally rotated, elbow flexed 90 degrees, and forearm in the neutral position. A total of three trials will be assessed on each side, with a rest break between trials. The average of three maximal force measurements per trial will be reported.
Change of the Capabilities of Upper Extremity Test (CUE-T) Scores | From baseline to the end of intervention at 2 weeks, post-intervention at 1 month, 2 months, and 3 months
  The Capabilities of Upper Extremity Test (CUE-T) will be used to evaluate the functional abilities, including 19 tasks (17 unilateral and 2 bilateral). Tasks involve a range of UE movements performed across proximal and distal joints for assessment of gross and fine motor function. Scoring for each item is based on ability to complete, rate of movement and time taken.

OTHER OUTCOMES:
Change of cortical excitability before and after intervention | From baseline to the post-intervention at 3 weeks
  Cortical excitability will be evaluated by measuring the amplitude of evoked motor potentials (MEP) elicited by transcranial magnetic stimulation (TMS). TMS will be delivered using a figure-of-eight coil (diameter 70 mm) attached to MagPro X30 stimulator (MagVenture, Mag2Health, Farum, Denmark). TMS-MEP from flexor carpi radialis (FCR) on the more-affected side will be recorded, since C5-C7 SCI typically impair active wrist flexion. The lowest intensity is defined as the resting motor threshold (RMT) and will be used as measures of cortical excitability. As an exploratory aim, the investigators will evaluate on a subset sample of each group (n=4).
Change of spinal excitability before and after intervention | From baseline to the post-intervention at 3 weeks
  Spinal excitability will be assessed by recording scTs-evoked MEPs. Monophasic scTS with 1-ms pulse width and an inter-stimuli interval of 5s will be applied to elicit MEPs by using the same current stimulator used in intervention. A peak-to-peak analysis will be performed in MATLAB (MathWorks Inc., Natick, MA, USA) software to evaluate the motor response and generate the sigmoid-shaped RC of scTS-MEP. Excitation threshold which indicates the excitability to the initial recruitment of motoneurons will be calculated. As an exploratory aim, the investigators will evaluate on a subset sample of each group (n=4).

CONTACTS AND LOCATIONS:
Overall Officials: Gail Forrest, PhD, Study Director — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Freitas RM, Sasaki A, Sayenko DG, Masugi Y, Nomura T, Nakazawa K, Milosevic M. Selectivity and excitability of upper-limb muscle activation during cervical transcutaneous spinal cord stimulation in humans. J Appl Physiol (1985). 2021 Aug 1;131(2):746-759. doi: 10.1152/japplphysiol.00132.2021. Epub 2021 Jun 17. PMID 34138648
- [Background] Gerasimenko YP, Lu DC, Modaber M, Zdunowski S, Gad P, Sayenko DG, Morikawa E, Haakana P, Ferguson AR, Roy RR, Edgerton VR. Noninvasive Reactivation of Motor Descending Control after Paralysis. J Neurotrauma. 2015 Dec 15;32(24):1968-80. doi: 10.1089/neu.2015.4008. Epub 2015 Aug 20. PMID 26077679
- [Background] Popovic MR, Kapadia N, Zivanovic V, Furlan JC, Craven BC, McGillivray C. Functional electrical stimulation therapy of voluntary grasping versus only conventional rehabilitation for patients with subacute incomplete tetraplegia: a randomized clinical trial. Neurorehabil Neural Repair. 2011 Jun;25(5):433-42. doi: 10.1177/1545968310392924. Epub 2011 Feb 8. PMID 21304020
- [Background] Kloosterman MG, Snoek GJ, Jannink MJ. Systematic review of the effects of exercise therapy on the upper extremity of patients with spinal-cord injury. Spinal Cord. 2009 Mar;47(3):196-203. doi: 10.1038/sc.2008.113. Epub 2008 Sep 30. PMID 18825160
- [Background] Burns AS, Marino RJ, Kalsi-Ryan S, Middleton JW, Tetreault LA, Dettori JR, Mihalovich KE, Fehlings MG. Type and Timing of Rehabilitation Following Acute and Subacute Spinal Cord Injury: A Systematic Review. Global Spine J. 2017 Sep;7(3 Suppl):175S-194S. doi: 10.1177/2192568217703084. Epub 2017 Sep 5. PMID 29164023
- [Background] Snoek GJ, IJzerman MJ, Hermens HJ, Maxwell D, Biering-Sorensen F. Survey of the needs of patients with spinal cord injury: impact and priority for improvement in hand function in tetraplegics. Spinal Cord. 2004 Sep;42(9):526-32. doi: 10.1038/sj.sc.3101638. PMID 15224087
- [Background] Zhang F, Momeni K, Ramanujam A, Ravi M, Carnahan J, Kirshblum S, Forrest GF. Cervical Spinal Cord Transcutaneous Stimulation Improves Upper Extremity and Hand Function in People With Complete Tetraplegia: A Case Study. IEEE Trans Neural Syst Rehabil Eng. 2020 Dec;28(12):3167-3174. doi: 10.1109/TNSRE.2020.3048592. Epub 2021 Jan 28. PMID 33382659
- [Background] Freyvert Y, Yong NA, Morikawa E, Zdunowski S, Sarino ME, Gerasimenko Y, Edgerton VR, Lu DC. Engaging cervical spinal circuitry with non-invasive spinal stimulation and buspirone to restore hand function in chronic motor complete patients. Sci Rep. 2018 Oct 19;8(1):15546. doi: 10.1038/s41598-018-33123-5. PMID 30341390
- [Background] Gad P, Lee S, Terrafranca N, Zhong H, Turner A, Gerasimenko Y, Edgerton VR. Non-Invasive Activation of Cervical Spinal Networks after Severe Paralysis. J Neurotrauma. 2018 Sep 15;35(18):2145-2158. doi: 10.1089/neu.2017.5461. PMID 29649928
- [Background] Inanici F, Samejima S, Gad P, Edgerton VR, Hofstetter CP, Moritz CT. Transcutaneous Electrical Spinal Stimulation Promotes Long-Term Recovery of Upper Extremity Function in Chronic Tetraplegia. IEEE Trans Neural Syst Rehabil Eng. 2018 Jun;26(6):1272-1278. doi: 10.1109/TNSRE.2018.2834339. PMID 29877852
- See also: Related Info — https://kesslerfoundation.org/research/studies/spinal-cord-transcutaneous-stimulation-upper-extremity-function-recovery-acute